CLINICAL TRIAL: NCT04822311
Title: Evaluating the Impact of Focused Muscle Contraction Therapy in Retired American Professional Football Players
Brief Title: Evaluating the Impact of Focused Muscle Contraction Therapy in Retire APF Players
Acronym: GH-APF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Responsible Party: Principal Investigator, Enrico Benedetti, Warren H. Cole Chair in Surgery, Professor and Head of Surgery, Medical Director, Abdominal Organ Transplant Program, University of Illinois at Chicago
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2019-0905
Record Dates: First submitted 2021-03-25; First posted 2021-03-30 (Actual); Last update posted 2023-06-09 (Actual); Status verified 2023-06

CONDITIONS: Chronic Pain Due to Injury; Acute Pain; Depression; Brain Injuries
MeSH Terms: conditions — Acute Pain; Depression; Brain Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Investigate the effects of an exercise intervention on retired APF players (Experimental): 20 retired APF players (≥ 18 years of age), who suffer from chronic pain, will be enrolled.
  Interventions: Behavioral: Experimental: Investigate the effects of an exercise intervention on retired APF players

INTERVENTIONS:
Behavioral: Experimental: Investigate the effects of an exercise intervention on retired APF players — Enrolled participants will perform a 18 months exercise intervention which involves 90 exercise rehabilitation training visits. In addition, participants will also be tested on various measures of health and function both at baseline (prior to intervention), at 6 months, 12 months, and 18 months (post intervention).

SUMMARY:
This study will investigate the effects of an exercise intervention on retired American professional football (APF) players. A total of 20 retired APF players (≥ 18 years of age), who suffer from chronic pain, will be enrolled. The study duration for each participants will be 18 months. Enrolled participants will perform a 18 months exercise intervention which involves 90 exercise rehabilitation training visits. In addition, participants will also be tested on various measures of health and function both at baseline (prior to intervention), at 6 months, 12 months, and 18 months (post intervention). All testing and result interpretation will be performed by trained research personnel. Participants are not University of Illinois at Chicago (UIC) participants; however, study testing visits will occur at UIC. All exercise intervention training visits will occur at Gh Fitlab.

DETAILED DESCRIPTION:
Methods:

Eligible participants will give voluntary informed consent to participate in the study. The study will include 20 retired APF players participating in a 18 month exercise rehabilitation. The study will consist of 94 visits (4 study testing visits and 90 exercise visits). Participants will come in for study testing visits at baseline (prior to starting the exercise program), at 6 months, at 12 months, and at 18 months(after ending the exercise program). Each of those visits will take about 2-3 hours. All testing done in the 4 test visits will help assess the participant's cardiovascular and functional responses and/or changes to the exercise intervention as indicated in the Objectives/Aims Section. The next section contains a list of the tests that will be performed at each visit. After the initial baseline visit, participants will come twice weekly, for roughly 1 hour each session, for 6 months (52 visits). From 6-12 months, participants will come once a week, for roughly 1 hour each session (26 additional visits). From 12-18 months, participants will come twice a month, for roughly 1 hour sessions (12 visits). All study testing visits will occur at the UIC. All exercise intervention training visits will occur at Gh Fitlab.

Study Testing Visits

If participants agree to be in the study, they will be asked to do the following procedures at baseline, 6 months, 12 months, and 18 months:

* participants will be asked to confirm their employment status each visit.
* participants height and weight will be measured and their body mass index (BMI) will be calculated. Additionally, we will measure body fat composition and lean body mass using a DEXA scan.
* We will ask about age, race, years in the APF league, number of concussions, number of fractures, surgical history, and list of pain medications.
* Waist circumference as well as blood pressure will be measured for general health markers.
* Participants exercise limit will be measured with a 1 Repetition Max test (1RM), a timed 8 foot walk down the hallway (if applicable), a timed sit to stand test (sitting and standing 5 times in a row-if applicable), maximum sit to stands, and a balance test (standing in 3 different positions for 10 seconds each). These three tests combine to form a score called a short performance battery score.
* Their strength and frailty will be measured using a grip dynamometer (squeezing a hand held device as hard as possible in their dominant hand three times.
* To evaluate general health, the PROMIS v.1.1 - Global Health questionnaire will be administered.
* To evaluate mental health and pain intensity, the PROMIS 29 Profile v2.0 will be administered.
* To evaluate quality of life, the SF-36 will be administered.
* To evaluate mental health, specifically depression, the Beck Depression Inventory will be administered.
* To evaluate brain anatomy and function, we will be using a quantitative EEG (QEEG), and a computer program called the Integrated Visual and Auditory Scale (IVA-2). For the QEEG, a technician will attach discs (electrodes) to the scalp of the participant using a special adhesive. Sometimes, an elastic cap fitted with electrodes is used instead. The electrodes are connected with wires to an instrument that amplifies the brain waves and records them on computer equipment. The electrodes don't transmit any sensations. They just record brain waves. For the IVA-2, you will perform tasks on a computer that will test sustained attention.
* To evaluate the measure of pain and disability, the Numeric Rating Scale and Pain Catastrophizing Scale will be administered.
* To evaluate fatigue, the Fatigue Severity Index will be administered.
* They will be asked to disclose the number of hospital visits they have had in the last 18 months.
* Their total weight lifted during their training session will also be recorded.

Exercise Training Visits

After the initial baseline visit, participants will begin their exercise training intervention which involves:

* Two days a week of exercise trainings for the first 6 months, and one day a week from 6-12 months. From 12-18 months, participants will then complete two days a month of exercise training. Each visit will last roughly one hour and will incorporate approximately 5-10 minute light warm-up plus stretching and then the exercises.
* At least twice weekly, GH Fitness staff will follow-up with participants via text message, email or a phone call to evaluate their physical progress and overall health and energy.
* On Weeks 6, 13, 18, 25, 41 and 52 participants will focus on cardio and endurance exercises. These exercises may include running in place, or using a recumbent (stationary) bike. All other weeks consist of basic strength training/resistance workouts.

ELIGIBILITY:
Inclusion Criteria:

* Retired APF player (there is no minimum duration or career length required no minimum duration or career length required)
* 18 years of age and older

Exclusion Criteria:

•This study will exclude non-English speaking participants as they would not be able to complete intensive survey requirement of the study as all surveys will be administered in the English language.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2019-10-24 (Actual); Primary Completion 2021-04-18 (Actual); Study Completion 2023-05-15 (Actual)

PRIMARY OUTCOMES:
Rate at which exercise will positively affect body composition | 18 months
  1. Exercise will positively affect body composition. With this hypothesis we will test whether muscle strength (dynamometer) and muscle mass (DEXA scan) changes after 6 months, 12 months, 18 months of an exercise intervention. Baseline measurement will be performed before the intervention, at 6 months, 12 months, and at the end of the study (18 months) with muscle mass measured by DEXA and strength measured again by dynamometer.

SECONDARY OUTCOMES:
Rate at which participants will see improvements in their physical abilities | 18 months
  2. We expect participants will see improvements in their physical abilities after 18 months in the exercise training sessions. This will be assessed by comparing baseline, 6 months, 12 months, and 18 months, 8 foot walk, timed sit to stand, and balance testing scores.
Rate at which participants will have overall improved sense of well-being, increased independence, quality of life, and decreased depression | 18 months
  3. Participants enrolled in the exercise intervention will have an overall improved sense of well-being, increased independence, quality of life, and decreased depression. Participants will be asked about their overall general health, mental health and pain intensity using the PROMIS, SF 36, BDI, Fatigue Severity Index, and pain assessments.
Rate at which participants will display alterations in brain wave function | 18 Months
  4. APF players with chronic pain described as greater than 5 out of a 10 point scale and lasting greater than 12 months, will display alterations in brain wave function consistent with abnormal function of the bilateral dorsolateral prefrontal cortex (DLPFC) , thalamus (relays motor and sensory signals to the cortex) , brainstem, primary somatosensory cortex (S1, postcentral gyrus of the anterior parietal lobe) and posterior parietal cortex (posterior to the primary somatosensory cortex)

CONTACTS AND LOCATIONS:
Overall Officials: Enrico Benedetti, MD, Principal Investigator — University of Illinois at Chicago
Locations (1):
- University of Illinois at Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2021-03-24): https://cdn.clinicaltrials.gov/large-docs/11/NCT04822311/Prot_000.pdf